CLINICAL TRIAL: NCT02671838
Title: Developing a Musculoskeletal Ultrasound Program as an Intervention to Improve Disease Modifying Anti-Rheumatic Drugs Adherence in Rheumatoid Arthritis: A Randomized Controlled Trial
Brief Title: A Musculoskeletal Ultrasound Program to Improve Disease Modifying Anti-Rheumatic Drugs Adherence in Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: US-01-2016
Record Dates: First submitted 2016-01-26; First posted 2016-02-02 (Estimated); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Musculoskeletal ultrasound program (Other): Participants will receive the musculoskeletal ultrasound program
  Interventions: Behavioral: Musculoskeletal ultrasound program
- Control (No Intervention): Participants will not be receiving the musculoskeletal ultrasound program.

INTERVENTIONS:
Behavioral: Musculoskeletal ultrasound program — Using a musculoskeletal ultrasound program to help improve medication adherence
  Arms: Musculoskeletal ultrasound program

SUMMARY:
Non-adherence to medications can lead to sub-optimal treatment in rheumatoid arthritis (RA) patients. In order to improve disease modifying anti-rheumatic drugs (DMARDs) adherence, the investigators are conducting a randomized controlled trial to test out an intervention to improve medications adherence among low adherers. This intervention involves the use of a musculoskeletal ultrasound program which allows RA patients to visualize their joint inflammation and damage real time while treatment adherence is simultaneously reinforced. In doing so, the investigators hope to improve patients' understanding of their joint disease and motivate the participants to adhere to their medications.

DETAILED DESCRIPTION:
This is a single center randomized controlled clinical trial conducted in the Singapore General Hospital. Eligible RA subjects meeting the inclusion and exclusion criteria will be screened using a medication adherence measure questionnaire. Thereafter 132 patients who are low adherers on the questionnaire will then be recruited and randomized (in a 1:1 ratio) to either (a) intervention arm (with musculoskeletal US program) or (b) control arm (without musculoskeletal US program), and followed up over a period of about 6 month.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients from 21 to 75 years old
* Underlying rheumatoid arthritis diagnosed using the 1987 or 2010 RA criteria
* On at least one of the following DMARDs (Methotrexate, Sulfasalazine, Hydroxychloroquine and/or Leflunomide)

Exclusion Criteria:

* Pregnancy

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Change in proportion of patients with a low adherence score using medication adherence measure (questionnaire) | baseline and 1 month

SECONDARY OUTCOMES:
Change in proportion of patients with a low adherence score using medication adherence measure (questionnaire) | baseline, 3 months and 6 months
Change in proportion of patients with a low adherence score using medication adherence measure (pharmacy dispense data) | baseline, 1 month, 3months and 6 months

OTHER OUTCOMES:
Change in clinical follow-up defaults (e.g. how often patients do not show up for their clinic appointments) | baseline, 3 months and 6 months
Change in clinical joint assessment outcomes(e.g. disease activity score 28) | baseline, 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tan, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No